CLINICAL TRIAL: NCT06224933
Title: Augmented Reality Real-Time Guidance for MRI-Guided Interventions
Brief Title: Augmented Reality For MRI-Guided Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Karun Sharma MD, Director of Interventional Radiology, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000648
Record Dates: First submitted 2023-11-22; First posted 2024-01-25 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Infections; Pain; Diagnosis
MeSH Terms: conditions — Infections; Pain; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients Undergoing Augmented Reality Image-Guided Needle Procedures (Experimental): Patients will undergo their standard of care image-guided needle biopsy, aspiration, or injection with the Augmented Reality system. Patients will be monitored for adverse events for two weeks following their procedure.
  Interventions: Device: Augmented Reality System

INTERVENTIONS:
Device: Augmented Reality System — Subjects will undergo image guided needle aspiration, injection, or biopsy facilitated by the Augmented Reality system. The Augmented Reality guidance system will be operated by the interventional radiologist in the MRI suite.

SUMMARY:
The purpose of this study is to determine feasibility and safety of using an augmented reality system in patients undergoing MRI-Guided needle procedures.

DETAILED DESCRIPTION:
This pilot clinical study is designed to evaluate the feasibility of using a needle guidance system during MRI-guided procedures in up to 12 patients. The MRI-compatible needle guidance system was developed under an NIH funded SBIR Phase II grant. This system has been evaluated by our Interventional Radiology team in phantom, volunteer, and cadaver studies which showed potential benefit of use in patients. Inclusion of the needle guidance system will not change the standard of care or substantively affect procedural technique as currently performed. This system provides the operator with an augmented reality (AR) display to better visualize the needle entry point and trajectory as it is inserted toward the target. This additional information could improve needle placement accuracy and shorten procedural time.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, ages 3 to 21
* Patient referred to Interventional Radiology for image-guided needle injection, aspiration, or biopsy.

Exclusion Criteria:

* Patients who are unable to give informed consent themselves or through their parents.
* Patients under 3 years of age
* Patients over 300 pounds.
* Patients who are claustrophobic and unable to tolerate MRI-guided procedure.
* Contraindications to MRI such as MR-unsafe implants.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-02-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility is measured by successful completion of greater than 80% of cases using the augmented reality needle guidance system. | 1 day
Safety of using the augmented reality needle guidance system will be evaluated through assessment of procedure related adverse events that occur within 7 days of the procedure. | 7 days

SECONDARY OUTCOMES:
Procedure time | 1 day
  Total procedure time.
Number of MRI scans | 1 day
  Number of MRI scans needed to complete the procedure, and size and depth of target will be recorded.
Clinical impressions of the system use and utility | 1 Day
  The operator will complete a usability form that captures ease of use using the Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Karun Sharma, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States